CLINICAL TRIAL: NCT06143787
Title: A Randomized, Double-blind, Multi-center, Placebo-controlled, Parallel-group Phase 3 Study to Compare the Efficacy, Acceptability, and Safety of Tranexamic Acid Oral Solution 5% With Placebo in the Prevention of Clinically Relevant Bleeding Events in Subjects Treated With Direct Oral Anticoagulants or Vitamin K Antagonists and Undergoing a Single or Multiple Tooth Extraction.
Brief Title: Effect of TXA Oral Sol 5% in Patients Treated With DOACs or VKA and Undergoing a Single or Multiple Tooth Extraction
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hyloris Developments (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HYL-P004-003; 2023-503719-13-00 (Other: EMEA)
Record Dates: First submitted 2023-11-15; First posted 2023-11-22 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2023-11

CONDITIONS: Bleeding From Teeth; Bleeding Prophylaxis
Keywords: bleeding teeth; Tranexamic Acid; Oral Solution; Tranexamic Acid Oral Solution 5%
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, multi-center, placebo-controlled, parallel-group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (T1) (Placebo Comparator): Standard hemostatic measures + Placebo matching with Tranexamic Acid Oral Solution 5%
  Interventions: Drug: Tranexamic acid
- Treatment (T2) (Experimental): Standard hemostatic measures + Tranexamic Acid Oral Solution 5%
  Interventions: Drug: Tranexamic acid

INTERVENTIONS:
Drug: Tranexamic acid — 7 days Oral rinsing following tooth extraction
  Other Names: Tranexamic Acid Oral Solution 5%

SUMMARY:
The purpose of this study is to assess the effect of Tranexamic Acid Oral Solution 5% in patients treated with direct oral anticoagulants or vitamin K antagonists and undergoing a single or multiple tooth extraction.

DETAILED DESCRIPTION:
The purpose of this study is to compare the efficacy, acceptability, and safety of Tranexamic Acid Oral Solution 5% with placebo in the prevention of clinically relevant bleeding events in subjects treated with direct oral anticoagulants or vitamin K antagonists and undergoing a single or multiple tooth extraction.

A total of approximately 280 subjects will be randomized in two equal treatment groups (approximately 140 subjects per group) to receive Tranexamic Acid Oral Solution 5% or placebo solution for 7 days. Following screening, eligible subjects can be randomized within 14 days when all eligibility criteria are confirmed. Randomized subjects will undergo tooth extraction(s) and treatment period. The treatment period ends at Visit 5 followed by the follow-up period. The maximal study duration is about 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Provide their signed study informed consent to participate.
2. Male or female ≥ 18 years of age at screening.
3. Body mass index (BMI) between 18.5 kg/m2 and 35 kg/m2, inclusively and body weight ≥ 50 kg.
4. Treated regularly for ≥ 3 months with direct oral anticoagu19lant (e.g., edoxaban, apixaban, rivaroxaban, dabigatran) or vitamin K antagonists (e.g., acenocoumarol, warfarin, etc.).
5. Subjects on VKAs can be enrolled if the subject's International Normalized Ratio (INR) at screening, but not more than 5 days before the dental extraction procedure is within the range of 2.0-3.5.
6. Subjects taking VKAs or DOACs can be enrolled if these are prescribed and used according to the approved product label.
7. Accepting to not discontinue his/her anticoagulant medication on the day of the extraction.
8. Scheduled to undergo a single or multiple (≤ 5 teeth, single-rooted, double-rooted, or multi-rooted, maximum 3 multi-rooted teeth and 2 different extraction sites) tooth extraction. Subjects with a single extraction site may have up to a maximum of 5 adjacent teeth extracted at the site, and subjects with two extraction sites may have up to a maximum of 3 adjacent extracted teeth at one site and 2 adjacent extracted teeth at the other site.
9. Considered as reasonably healthy to follow the study procedures as documented by the medical history, physical examination, and vital sign assessments.
10. Subjects with a platelet count of 100,000-500,000 (inclusive) platelets per microliter.
11. Subject with hemoglobin ≥ 12.0 g/dL (male) or ≥ 11.0 g/dL (female).
12. Willing to avoid alcohol consumption for the duration of the study.
13. Willing and able to adhere to the study assessment schedule and other protocol requirements as evidenced by a written informed consent.
14. Negative pregnancy test in females of childbearing potential at Screening and Day 1 visit.
15. Women must be post-menopausal (defined as no menses for 12 months without an alternative medical cause), surgically sterile, or willing to use highly effective method of birth control which is defined as those which result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly (refer to Table 4 in protocol Section 8.2.11 for further information on acceptable and unacceptable birth control methods). The Investigator is responsible for determining whether the subject has adequate birth control for study participation.

Exclusion Criteria:

1. Any coagulation disorders requiring TXA.
2. Wisdom teeth extraction.
3. History of severe allergy or allergic reactions or hypersensitivity to the study drug or any component of its formulations or related drugs or heparin
4. Subjects with type IV periodontitis (as per American Dental Association Classification) (see Appendix 1).
5. History of subarachnoid hemorrhage.
6. Active intravascular clotting (defined as a history of thrombosis within the past 3 months).
7. Blood in the urine (macroscopic hematuria) at Screening.
8. Renal function test result of estimated glomerular filtration rate ≤ 15 mL/min/1.73 m² at Screening.
9. Any ongoing or planned dual anti-platelet treatment for the duration of subject's participation in the study (any 2 of the following: aspirin, dipyridamole, or any thienopyridine, i.e., clopidogrel, prasugrel, ticlopidine, ticagrelor). However, subjects receiving a very low dose aspirin (≤ 160 mg) may be enrolled.
10. Any ongoing or planned oncological treatment for the duration of subject's participation in the study.
11. Any immunocompromising condition.
12. Use of any recreational drugs or history of drug addiction.
13. Positive alcohol breath test at Screening and Day 1.
14. Participating in any other clinical study or has received treatment with any investigational drug or device within 3 months prior to screening.
15. History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of the investigational drug, might affect interpretation of the results of the study, or renders the subject at high risk for treatment complications (including but not limited to diseases such as uncontrolled diabetes, any haemato-oncological condition [e.g., leukemia], any congenital hematological condition [e.g., hemophilia]).
16. Severe uncontrolled arterial hypertension, e.g., > 200 mmHg systolic or > 110 mmHg diastolic blood pressure at two consecutive readings.
17. Subjects who are found positive to human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) serological tests.
18. Use of hormonal methods of birth control that increase the risk of thrombosis (e.g., estrogen-containing contraceptives). Refer to Table 4 in protocol Section 8.2.11 for further information on acceptable and unacceptable birth control methods.
19. Women with intended pregnancy or breast-feeding.
20. Planned soft (other than extraction site) or hard oral tissue biopsy on the day of the surgery.
21. Subjects who are evaluated to have a negative risk-benefit ratio to participate in this study (e.g., high risk of severe bleeding).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2024-12-27 (Estimated); Study Completion 2024-12-27 (Estimated)

PRIMARY OUTCOMES:
Number of clinically relevant postoperative oral bleeding episodes | 7 days
  Number of clinically relevant postoperative oral bleeding episodes (including clinically relevant orofacial hematomas)

SECONDARY OUTCOMES:
Number of postoperative oral bleeding episodes | 7 days
  Number of postoperative oral bleeding episodes (including clinically relevant and not clinically relevant bleedings and orofacial hematomas)
Number of delayed postoperative oral bleeding episodes | 7 days
  Number of delayed postoperative oral bleeding episodes, both clinically relevant and not clinically relevant, in all subjects.
Number of early postoperative oral bleeding episodes | 7 days
  Number of early (less than 24 h post-tooth extraction) postoperative oral bleeding episodes, both clinically relevant and not clinically relevant, in all subjects
Perioperative and immediate post-operative duration | 7 days
  Perioperative and immediate post-operative (procedural bleeding) duration (min, all types of oral bleeding).
Medication Acceptability Questionnaire (MAQ) completed | 7 days
  Medication Acceptability Questionnaire (MAQ) for Tranexamic Acid Oral Solution 5% use completed in all subjects

CONTACTS AND LOCATIONS:
Overall Officials: Todd Bertoch, Dr., Principal Investigator — JBR Clinical Research (CenExcel)
Locations (19):
- United States (4):
  - Loma Linda University School of Dentistry, Loma Linda, California
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - JBR Clinical Research (CenExel), Millcreek, Utah
  - Roseman University of Health Sciences, College of Dental Medicine, South Jordan, Utah
- Croatia (4):
  - Clinical Hospital Center Rijeka, Dental clinic, Rijeka
  - University Hospital of Split Department of Oral surgery, Split
  - Dental Clinic Zagreb, Zagreb
  - University hospital Dubrava Department of oral surgery, Zagreb
- Hungary (3):
  - Semmelweis Egyetem, Fogorvostudományi Kar, Arc-Állcsont-Szájsebészeti És Fogászati Klinika, Budapest
  - SZTE SZAKK Arc-, Állcsont- és Szájsebészeti Klinika, Szeged
  - Arc-, Állcsont-, Szájsebészeti Osztály, Veszprém
- Romania (3):
  - "Dr. Carol Davila" Central Military Emergency University Hospital Bucharest, Bucharest
  - Trident Clinic, Bucharest
  - SCJU Craiova, Craiova
- Spain (5):
  - Medicine and Healthcare Science Faculty of Barcelona University (Campus Bellvitge, Barcelona
  - Puerta del Mar University Hospital, Cadiz
  - Jerez Center Health Center, Jerez de la Frontera
  - Hospital Universitario La Paz, Madrid
  - Institute of Biotechnology of Seville (IBIS), Seville